CLINICAL TRIAL: NCT00602537
Title: Treatment of Bipolar Type II Major Depression
Brief Title: Antidepressant Therapy in Treating Bipolar Type II Major Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01MH060353-02 (NIH); R01MH060353-02 (NIH); 2R01MH060353-06A2 (NIH)
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Bipolar Disorder; Depression
Keywords: Bipolar Type II Disorder; Hypomania; Antidepressant; Mood Stabilizer; Venlafaxine; Lithium Carbonate; Major Depressive Episode; Hypomanic Episodes; Prevention of Depression Relapse
MeSH Terms: conditions — Bipolar Disorder; Depression; Mania | interventions — Venlafaxine Hydrochloride; Lithium Carbonate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Experimental): Antidepressant therapy
  Interventions: Drug: Venlafaxine
- II (Active Comparator): Mood stabilizer therapy
  Interventions: Drug: Lithium Carbonate

INTERVENTIONS:
Drug: Venlafaxine — 75 to 375 mg
  Arms: I
Drug: Lithium Carbonate — 300 to 2400 mg
  Arms: II

SUMMARY:
This study will compare the safety and effectiveness of antidepressant therapy versus mood stabilizing therapy in treating people with bipolar type II major depression.

DETAILED DESCRIPTION:
Bipolar type II (BP II) depression affects 2.5% of the U.S. adult population. People with BP II disorder do not experience the manic episodes that are characteristic of BP I disorder, but rather they experience more modest mood swings with a greater number of major depressive episodes (MDEs). These MDEs are associated with high rates of disease and death. The treatment of BP II depression remains a challenge for clinicians. Mood stabilizer (MS) monotherapy is the current recommended treatment for BD II MDE, but there is reason to believe that antidepressant drug (AD) monotherapy could also be an effective treatment. However, concerns over AD-induced manic switch episodes have limited the use of this treatment option. Preliminary studies using the ADs fluoxetine or venlafaxine have shown success in treating and lowering the manic switch rate of those with BP II MDE. This study will compare the safety and effectiveness of AD monotherapy versus MS monotherapy in treating people with BP II major depression.

Participation in this double-blind study will last up to 9 months. After screening, which includes a medical and psychiatric history review, a physical exam, an electrocardiogram (EKG) test, clinical laboratory tests, a urine-based drug test, and a pregnancy test if applicable, participants will be randomly placed into one of two treatment groups. Participants in the AD monotherapy group will be treated with venlafaxine, and participants in the MS monotherapy group will be treated with lithium. During the first 12 weeks, there will be a total of nine study visits lasting between 45 and 60 minutes. In these visits, participants will receive their study drug and will undergo various assessments, including a review of medication history and side effects, vital sign measurements, and questionnaires about depression and daily functioning. Blood samples will be taken at most visits.

Participants who respond well during the initial 12 weeks of therapy with either drug will have the option to continue treatment for 6 additional months. During this time, participants will continue their assigned treatment and will attend five monthly study visits that will repeat previous assessments and procedures.

For information on a related study, please follow this link:

http://clinicaltrials.gov/show/NCT00044616

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for Axis I bipolar II disorder
* Meets DSM-IV criteria for Axis I major depressive episode
* Score of 16 on 17-item HAM-D rating scale
* Not taking monoamine oxidase inhibitors (MAOI) for more than 2 weeks prior to study entry
* Willing to use an effective form of birth control throughout the study

Exclusion Criteria:

* History of mania
* Current primary Axis I diagnosis other than bipolar II disorder
* Alcohol or drug dependence within 3 months prior to study entry
* Contraindication to treatment with venlafaxine or lithium
* Unstable medical condition (e.g., thyroid disease, hypertension, or angina pectoris)
* Pregnant or breastfeeding
* Experiencing suicidal thoughts
* Requires hospitalization
* Requires concurrent neuroleptic or MS therapy
* Requires concurrent AD therapy
* Current psychotic features
* Inadequate trial of therapy at the time of initial screening visit
* History of intolerance to either venlafaxine or lithium
* Unlikely to participate in a 36-week trial
* Presence of apparent secondary gain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2007-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. DeRubeis, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Depression Research Unit - University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lorenzo-Luaces L, Amsterdam JD, DeRubeis RJ. Residual anxiety may be associated with depressive relapse during continuation therapy of bipolar II depression. J Affect Disord. 2018 Feb;227:379-383. doi: 10.1016/j.jad.2017.11.028. Epub 2017 Nov 8. PMID 29149756
- [Derived] Lorenzo-Luaces L, Amsterdam JD. Effects of venlafaxine versus lithium monotherapy on quality of life in bipolar II major depressive disorder: Findings from a double-blind randomized controlled trial. Psychiatry Res. 2018 Jan;259:455-459. doi: 10.1016/j.psychres.2017.11.025. Epub 2017 Nov 8. PMID 29136600
- [Derived] Amsterdam JD, Lorenzo-Luaces L, DeRubeis RJ. Comparison of treatment outcome using two definitions of rapid cycling in subjects with bipolar II disorder. Bipolar Disord. 2017 Feb;19(1):6-12. doi: 10.1111/bdi.12462. Epub 2017 Feb 3. PMID 28160351
- [Derived] Amsterdam JD, Lorenzo-Luaces L, DeRubeis RJ. Step-wise loss of antidepressant effectiveness with repeated antidepressant trials in bipolar II depression. Bipolar Disord. 2016 Nov;18(7):563-570. doi: 10.1111/bdi.12442. Epub 2016 Nov 2. PMID 27805299
- [Derived] Amsterdam JD, Lorenzo-Luaces L, Soeller I, Li SQ, Mao JJ, DeRubeis RJ. Short-term venlafaxine v. lithium monotherapy for bipolar type II major depressive episodes: effectiveness and mood conversion rate. Br J Psychiatry. 2016 Apr;208(4):359-65. doi: 10.1192/bjp.bp.115.169375. Epub 2016 Feb 18. PMID 26892848
- [Derived] Lorenzo-Luaces L, Amsterdam JD, Soeller I, DeRubeis RJ. Rapid versus non-rapid cycling bipolar II depression: response to venlafaxine and lithium and hypomanic risk. Acta Psychiatr Scand. 2016 Jun;133(6):459-69. doi: 10.1111/acps.12557. Epub 2016 Jan 24. PMID 26803764
- [Derived] Amsterdam JD, Lorenzo-Luaces L, Soeller I, Li SQ, Mao JJ, DeRubeis RJ. Safety and effectiveness of continuation antidepressant versus mood stabilizer monotherapy for relapse-prevention of bipolar II depression: A randomized, double-blind, parallel-group, prospective study. J Affect Disord. 2015 Oct 1;185:31-7. doi: 10.1016/j.jad.2015.05.070. Epub 2015 Jun 26. PMID 26143402

RESULTS

PARTICIPANT FLOW:
Groups:
- Antidepressant Therapy: Venlafaxine: 75 to 375 mg
- Mood Stabilizer Therapy: Lithium Carbonate: 300 to 2400 mg
Period: 12 Week Double Blind Comparison
Arm/Group | Antidepressant Therapy | Mood Stabilizer Therapy
Started | 65 | 64
Responded | 44 | 22
Completed | 42 | 17
Not Completed | 23 | 47
Not completed — Adverse Event | 2 | 5
Not completed — Lack of Efficacy | 13 | 23
Not completed — Lost to Follow-up | 5 | 6
Not completed — Withdrawal by Subject | 3 | 13
Period: Follow Up Study Comparison
Arm/Group | Antidepressant Therapy | Mood Stabilizer Therapy
Started | 42 | 17
Completed | 31 | 14
Not Completed | 11 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 8 | 1
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Antidepressant Therapy | Mood Stabilizer Therapy | Total
Number analyzed (Participants) | 42 | 17 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (11.4) | 43.1 (15.2) | 42.2 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 8 | 32
  Male | 18 | 9 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 37 | 12 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Inter-episode recovery [Count of Participants; unit: Participants] | 14 | 2 | 16
Age 1st major depressive episode [Mean (Standard Deviation); unit: years] | 19.0 (7.7) | 17.4 (5.4) | 18.5 (7.1)
Age 1st hypomanic episode [Mean (Standard Deviation); unit: years] | 20.7 (7.6) | 16.2 (10.0) | 19.4 (8.5)
Number of lifetime major depressive episodes [Mean (Standard Deviation); unit: Episodes] | 28.4 (50.4) | 33.3 (49.7) | 29.9 (11.0)
Number of lifetime hypomanic episodes [Mean (Standard Deviation); unit: Episodes] | 45.8 (66.4) | 32.2 (47.3) | 41.9 (61.4)
Baseline HRSD score [Mean (Standard Deviation); unit: units on a scale] — This scale refers to the 17-item Hamilton Rating Scale for Depression and measures patient depressive severity. The scale ranges from 0 to 52, with higher scores representing worse outcome.
  units on a scale | 19.4 (3.6) | 18.8 (3.3) | 19.2 (3.5)
Baseline YMRS score [Mean (Standard Deviation); unit: units on a scale] — This scale refers to the Young Mania Rating Scale and measures manic symptoms. The scale ranges from a minimum score of 0 to a maximum score of 60, with higher scores representing worse outcome.
  units on a scale | 0.8 (1.7) | 0.6 (1.4) | 0.8 (1.6)
Duration major depressive episode [Median (Full Range); unit: months] | 4.5 [.75 to 60] | 4.0 [0 to 396] | 4 [0 to 60]
Baseline HRSD Score for Follow-Up study [Mean (Standard Deviation); unit: units on a scale] — This scale refers to the 17-item Hamilton Rating Scale for Depression and measures patient depressive severity. The scale ranges from 0 to 52, with higher scores representing worse outcome.
  units on a scale | 4.3 (2.8) | 4.4 (3.4) | 4.3 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Depressive Relapse
Description: These subjects must be responders. Outcome measures were obtained at continuation weeks. Participant would be considered "depressive relapse" if relapsed by any of these times.
Time Frame: Weeks 16, 20, 24, 30, 36
Measure: Count of Participants; unit: Participants
Arm/Group | Antidepressant Therapy | Mood Stabilizer Therapy
Number analyzed (Participants) | 40 | 15
Participants | 3 | 4

2. Secondary Outcome: Treatment-Emergent Mood Symptoms
Description: These subjects must be responders.
Time Frame: Measured at Weeks 12 and 36
Measure: Count of Participants; unit: Participants
Arm/Group | Antidepressant Therapy | Mood Stabilizer Therapy
Number analyzed (Participants) | 40 | 15
Participants
  Any depression | 15 | 11
  Any subsyndromal hypomania | 3 | 3

ADVERSE EVENTS:
Arm/Group | Antidepressant Therapy | Mood Stabilizer Therapy
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/64
Other Adverse Events (participants affected / at risk) | 0/65 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No